CLINICAL TRIAL: NCT06426797
Title: Safety and Efficacy of Cadonilimab Combined With Anlotinib in Neoadjuvant Treatment of Locally Advanced Resectable Esophageal Squamous Cell Carcinoma: a Single Arm, Phase II Study
Brief Title: Neoadjuvant Cadonilimab Combined With Anlotinib in Locally Advanced Resectable Esophageal Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Akeso Pharmaceuticals, Inc. (Other)
Responsible Party: Principal Investigator, Yang Fan, MD, Professor of Thoracic Surgery, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-IIT-C-N1-0104
Record Dates: First submitted 2024-05-19; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Locally Advanced Esophageal Squamous Cell Carcinoma
Keywords: esophageal squamous cell carcinoma; neoadjuvant immunotherapy; pathological complete response
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — anlotinib

STUDY DESIGN:
Intervention Model Description: Patients with locally advanced resectable esophageal squamous cell carcinoma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- locally advanced ESCC (Experimental): Patients with locally advanced esophageal squamous cell carcinoma
  Interventions: Drug: Cadonilimab plus anlotinib

INTERVENTIONS:
Drug: Cadonilimab plus anlotinib — cadonilimab (10mg/Kg, ivgtt, d1) and anlotinib (12mg, P.O., d1-d14) on a 21-day regimen for 3 cycles

SUMMARY:
The goal of this clinical trial is to learn if cadonilimab combined with anlotinib can be a safe and effective neoadjuvant therapy in patients with locally advanced resectable esophageal squamous cell carcinoma (ESCC). The main questions it aims to answer are:

What level of pathological complete response (pCR) rate can be achieved with this neoadjuvant regimen? Is this neoadjuvant regimen safe enough with acceptable toxicity?

Participants will:

Receive cadonilimab (10mg/Kg, ivgtt, d1) and anlotinib (12mg, P.O., d1-d14) on a 21-day regimen for 3 cycles.

Undertake radical resection of ESCC after neoadjuvant therapy if there is no surgical contraindication.

Accept an follow-up for 2 years after surgery.

DETAILED DESCRIPTION:
Esophageal cancer has a high incidence in China, among which esophageal squamous cell carcinoma is the most common. Neoadjuvant chemoradiotherapy combined with surgery is currently the recommended treatment modality for locally advanced esophageal cancer, but the side effects of chemoradiotherapy are serious, which increases the risk of surgery.

Immune checkpoint inhibitors have made significant progress in the field of cancer treatment in recent years, and have now become an important treatment method for advanced and metastatic esophageal cancer. Several trials on neoadjuvant immuno-chemotherapy demonstrated better outcomes with acceptable toxicity compared to traditional chemoradiotherapy. Cadonilimab is a dual immune antibody drug comprised of PD-1 antibody and CTLA-4 antibody, which has the anti-tumor effect of two immune checkpoint pathways at the same time.

On the other hand, angiogenesis plays a vital role in the growth and metastasis of tumors, and anti-angiogenic drugs have become an important part of cancer treatment. Anlotinib is an oral, small molecule anti-angiogenic targeted agent that has been approved for use in a variety of cancer treatments.

This study plans to conduct a prospective study of cadonilimab combined with anlotinib in the neoadjuvant treatment of resectable esophageal squamous cell carcinoma, and aims to explore the efficacy and safety of this neoadjuvant regimen that avoids chemoradiotherapy in locally advanced resectable esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent and understand and agree to comply with the requirements of this study as well as the assessment schedule.
2. Be at least 18 years of age on the date of signing the ICF.
3. Histopathologically confirmed esophageal squamous cell carcinoma: the clinical stage is T1-2N1-3M0, T2 (diameter≥3 cm) N0M0 or T3-4aN0-3M0 (stage II-IVA), and the staging should be based on the AJCC 8th edition esophageal cancer staging system.
4. Patients are asked to provide an archival tumor tissue sample (FFPE tissue block or approximately 15 [≥6] freshly cut unstained FFPE sections) and a pathology report of this baseline sample. If no archival sample is available or the sample is not available, a biopsy sample is requested at baseline.
5. Prior to study enrollment, patients are evaluated by thoracic surgeon in charge of surgery to verify that they meet the study requirements for R0 resection with radical curative intent.
6. Cardiac and pulmonary function is good, and surgical resection for curative purposes is confirmed, and cardiopulmonary function tests and respiratory or cardiology consultation can be completed if necessary.
7. Measurable disease as assessed by the investigator according to RECIST version 1.1.
8. Eligible for anlotinib treatment.
9. ECOG performance status ≤ 2 points.
10. ≤ 14 days prior to enrollment, the following laboratory test values during the screening period suggest that the patient has good organ function:

    * Patient has not had a blood transfusion or use of growth factor supportive therapy within ≤14 days prior to blood draw, when the following items are tested prior to enrollment:

      * Absolute neutrophil count ≥ 1.5 x 109/L
      * Platelet ≥ 75×109/L
      * Hemoglobin ≥ 90 g/L
    * Glomerular filtration rate (GFR) estimated by the Cooperative Equation for Epidemiology of Chronic Kidney Disease ≥45mL/min/1.73 m2.
    * Serum total bilirubin ≤ 1.5 × upper limit of normal (ULN) (total bilirubin must be <3 ×ULN in patients with Gilbert's syndrome).
    * AST and ALT≤2.5 ×ULN.
    * Patients not receiving anticoagulant therapy: International normalized ratio or activated partial prothrombin time ≤ 1.5× ULN.
11. Females of childbearing potential must be willing to practice highly effective contraception for the duration of the study, and for ≥120 days after the last dose of cadonilimab or anlotinib, whichever occurs later, and have a negative urine or serum pregnancy test result within ≤7 days prior to enrollment.

Exclusion Criteria:

1. Previous treatment for current esophageal cancer, including chemotherapy or radiotherapy.
2. Prior receipt of antibodies or drugs targeting immune checkpoint pathways, including but not limited to anti-cytotoxic T-lymphocyte-associated antigen-4 (anti-CTLA-4), anti-PD-1, and anti-PD-L1 therapeutic antibodies.
3. Patients with non-squamous cell carcinoma.
4. Presence of locally advanced, unresectable disease, regardless of disease stage and presence or absence of metastases (stage IV).
5. Active autoimmune disease or history of autoimmune disease that may recur.

   Note: Patients with the following conditions do not need to be excluded and can proceed for further enrollment screening:
   * Well-controlled type I diabetes
   * Hypothyroidism (as long as it is treated with hormone replacement therapy alone)
   * Well-controlled celiac disease
   * Skin conditions that do not require systemic treatment (e.g., vitiligo, psoriasis, alopecia)
   * Any other illness that is not expected to recur in the absence of an external trigger
6. Any active malignancy in the ≤ 2 years prior to enrollment, with the exception of the specific cancers studied in this study and cancers that have recured locally after radical therapy (e.g., resected basal cell or squamous cell skin cancer, superficial bladder cancer, cervical or breast carcinoma in situ).
7. Any condition requiring systemic treatment with corticosteroids (prednisone or equivalent> 10 mg/day) or other immunosuppressive medications within ≤14 days prior to enrollment.

   Note: Patients with current or prior use of any of the following steroid regimens do not need to be excluded:
   * Adrenal replacement steroids (prednisone or equivalent> 10 mg/day)
   * Topical, ocular, intra-articular, intranasal, or inhaled corticosteroids with very low systemic absorption
   * Short-term (≤7 days) prophylactic use of corticosteroids (e.g., contrast allergy) or for the treatment of non-autoimmune diseases (e.g., delayed-type hypersensitivity reactions caused by contact allergens)
8. Poorly controlled diabetes mellitus ≤ 14 days prior to enrollment, or abnormal laboratory test results of potassium, sodium, or corrected calcium > grade 1 (regardless of standard medical management) or ≥ grade 3 hypoalbuminemia.
9. Has a history of interstitial lung disease, non-infectious pneumonitis, or poorly controlled diseases, including pulmonary fibrosis, acute lung disease, etc.
10. Severe chronic or active infection requiring systemic antibacterial, antifungal or antiviral therapy, including tuberculosis infection, etc. Severe infection within 4 weeks prior to enrollment, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia.
11. Known history of HIV virus infection.
12. Patients with untreated chronic hepatitis B or HBV carriers with hepatitis B virus (HBV) DNA ≥ 500 IU/mL, or patients with active hepatitis C virus (HCV) should be excluded.

    Note: Patients with inactive hepatitis B surface antigen (HBsAg) carriers, treated and stable hepatitis B carriers (HBV DNA < 500 IU/mL), and cured hepatitis C patients can be enrolled.
13. Any major surgical procedure requiring general anesthesia ≤ 28 days prior to enrollment.
14. Previous allogeneic stem cell transplantation or organ transplantation.
15. Any of the following cardiovascular risk factors:

    * Cardiogenic chest pain within 28 days prior to enrollment, defined as moderate pain with instrumental limitation of activities of daily living.
    * Symptomatic pulmonary embolism within 28 days prior to enrollment.
    * Any history of acute myocardial infarction within 6 months prior to enrollment.
    * Any history of heart failure consistent with New York Heart Association Classification Class III or IV≤ 6 months prior to enrollment.
    * Any ≥ grade 2 ventricular arrhythmic event within 6 months prior to enrollment (inclusive).
    * Any history of cerebrovascular accident within 6 months prior to enrollment.
    * Hypertension that remains uncontrolled with standard antihypertensive medication within 28 days prior to enrollment.
    * Syncope or seizures ≤ 28 days prior to enrollment.
16. History of severe allergic reaction to chimeric or humanized antibodies or fusion proteins.
17. Received any other chemotherapy, immunotherapy (e.g., interleukin, interferon, thymosin), or any investigational therapy during the study period.
18. Patients who have not returned to baseline or stable levels of toxic side effects (due to prior antineoplastic therapy) unless the AE is not considered to pose a safety risk (e.g., alopecia, neuropathy, and specific laboratory abnormalities).
19. Received a live vaccine ≤ 4 weeks prior to enrollment. Note: Seasonal influenza vaccines are usually inactivated and are therefore permitted. Intranasal vaccination is a live vaccine, so it is not allowed.
20. Has an underlying medical condition (including laboratory abnormalities) or alcohol/drug abuse or dependence that, in the opinion of the investigator, is detrimental to study drug administration or affects the interpretation of drug toxicity or adverse events, or in the judgment of the investigator that the patient's adherence during the study is not adequate that could affect compliance.
21. Participating in another therapeutic clinical study at the same time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) Rate | Within 1 week after surgery
  Pathological complete response (pCR) rate is defined as the percentage of participants with no residual viable tumor in primary tumor site or lymph nodes as evaluated by blinded independent pathological review (BIPR).

SECONDARY OUTCOMES:
Major Pathological Response (MPR) Rate | Within 1 week after surgery
  Major pathological response (MPR) rate is defined as the percentage of participants with less than or equal to 10% of residual viable tumor in primary tumor site or lymph nodes as evaluated by blinded independent pathological review (BIPR). Viable tumors in situ carcinoma should not be included in MPR calculation.
Objective Response Rate (ORR) | Within 1 week before surgery
  Objective response rate (ORR) is defined as the Percentage of participants achieving complete response (CR) or partial response (PR) in all patients with measurable disease at baseline, as assessed by the investigator according to RECIST version 1.1.
Treatment Emergent Adverse Events (TEAE) | Up to 24 months after participation
  The incidence and severity of treatment emergent adverse events (including adverse events, serious adverse events and immune-related adverse events) among all participants.
Event-free Survival (EFS) | Up to 24 months after participation
  EFS is defined as the time from participation to any of the following events: progression of disease, recurrence disease, or death due to any cause. Progression/recurrence will be assessed either by biopsy assessed by local pathologist or by investigator-assessed imaging using RECIST version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Fan Yang, M.D., Study Chair — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No